CLINICAL TRIAL: NCT07009912
Title: A Single-arm, Monocentric, Cross-sectional, Pilot Study Evaluating Updated Features for The ROSA® Knee System, v1.5, in Patients Undergoing Primary Total Knee Arthroplasty
Brief Title: ROSA® Knee System V1.5 Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCA2025-20TDS
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Knee Arthroplasty, Total; Robotic Surgical Procedures; Joint Diseases; Knee Osteoarthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Single-arm, monocentric, cross-sectional, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Zimmer Biomet ROSA® Knee System, v1.5 (Experimental): This study will include a single-arm of patients who qualify for robotic-assisted (RA) total knee arthroplasty (TKA) with the ROSA® Knee System and are planned to receive commercially available and compatible implants.
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Robotic-assisted primary total knee arthroplasty, evaluating updated features for the Zimmer Biomet ROSA® Knee System, v1.5.

SUMMARY:
This pilot study seeks to evaluate the initial safety and usability of new features for the ROSA® Knee System, v1.5 and plan design modifications as needed.

The primary objectives will be assessed by measuring:

1. Intra-operative complications
2. Verification that the device performs as intended
3. Overall surgeon satisfaction with the instrumentation.

DETAILED DESCRIPTION:
This study will involve single-arm, monocentric, cross-sectional observations conducted on the day of surgery. All assessments will take place during the pre-operative, intra-operative, and immediate postop periods on the day of surgery, with no additional follow-up beyond the procedure as robotic-assisted surgery using the current version of the robot is part of routine practice.

The safety of the system is the primary endpoint. This will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The secondary endpoint is defined by the usability of Zimmer Biomet ROSA® Knee System, v1.5. It will be assessed by:

1. Robotic log files to assess differences in the proposed plans by the system's new features and plan approved by the surgeon, along with time spent in the planning panel.
2. Surgeon satisfaction with the new features.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years of age
* Independent of study participation, patient is a candidate for primary total knee arthroplasty using commercially available and compatible implants in accordance with product labeling
* Patient is willing and able to provide written Informed Consent by signing and dating the EC approved Informed Consent form

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Procedure-Emergent Adverse Events, to assess the Safety of the ROSA® Knee System v1.5 System | Intra-operative observations, with immediate post-operative documentation and reporting period.
  The safety of the system will be assessed by monitoring the frequency and incidence of adverse events.
  This will occur through the reporting of adverse events that outline the details and relationship to:
  1. Device
  2. Procedure
  3. Instruments
  4. Cement in order to determine device-related or non-device-related complications that occur during the procedure. Thus the incidence of procedure-emergent adverse events will notify and quantify the safety of the features added to the subject device (ROSA® Knee System v1.5 System)

SECONDARY OUTCOMES:
Verification and Usability of the OptimiZe Planning and Activ Track Investigational Features of the ROSA® Knee System v1.5 System | Intra-operative evaluation, with immediate post-operative assessment and documentation. Data and statistical analysis will take place after the recruitment period has concluded.
  Robotic log files will be evaluated to assess the following:
  a) The delta between the OptimiZe proposed plan and the final plan approved by the surgeon, planned and final laxities, planned and final resections thus allowing for conclusions to be drawn from objective datapoints on the verification of the OptimiZe planning feature, and its validation to execute the proposed plan.
  Additionally, surgeon satisfaction with the features will be evaluated with the following questionnaire (Case Report Form), to determine usability:
  1. Were you able to perform tracker calibration?
  2. Were you able to complete painting?
  3. Were you able to perform the contact point step?
  4. Overall, how satisfied are you with the usability of OptimiZe to assist with planning?
  5. Overall, how satisfied are you with the usability of Activ Track to complete the resections?
  6. How likely are you to recommend The ROSA Knee System v1.5 application to a peer? Q1-4 are yes/no, Q5-6 are subjective scales with 5 answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Kensington Private Hospital, Kensington, Whangarei, New Zealand

IPD SHARING:
Plan to Share IPD: No